CLINICAL TRIAL: NCT06742190
Title: A Phase 3, Randomized, Double-Blinded, Double-Dummy Study Evaluating the Efficacy and Safety of Empasiprubart Versus Intravenous Immunoglobulin in Adults With Multifocal Motor Neuropathy
Brief Title: A Study to Assess the Efficacy and Safety of Empasiprubart Versus IVIg in Adults With Multifocal Motor Neuropathy
Acronym: Empassion
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-117-2302; 2024-516473-72-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Multifocal Motor Neuropathy (MMN); MMN
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - empasiprubart + IVIg-placebo (Experimental): During the double blinded - double dummy part A, participants receive empasiprubart and a placebo resembling the IVIg treatment in this arm
  Interventions: Biological: Empasiprubart; Other: IVIg-placebo
- Part A - IVIg + empasiprubart-placebo (Active Comparator): During the double blinded - double dummy part A, participants receive IVIg and a placebo resembling the empasiprubart treatment in this arm
  Interventions: Biological: IVIG (Intravenous Immunoglobulin); Other: Empasiprubart-placebo
- Part B - empasiprubart (Experimental): After completion of part A, participants can proceed to part B where they receive empasiprubart (no IVIg)
  Interventions: Biological: Empasiprubart

INTERVENTIONS:
Biological: Empasiprubart — Intravenous infusion of empasiprubart
  Arms: Part A - empasiprubart + IVIg-placebo; Part B - empasiprubart
Biological: IVIG (Intravenous Immunoglobulin) — Intravenous infusion of IVIg
  Arms: Part A - IVIg + empasiprubart-placebo
Other: Empasiprubart-placebo — A placebo resembling the empasiprubart treatment
  Arms: Part A - IVIg + empasiprubart-placebo
Other: IVIg-placebo — A placebo resembling the IVIg treatment
  Arms: Part A - empasiprubart + IVIg-placebo

SUMMARY:
The main purpose of this study is to compare empasiprubart and IVIg in adult patients with MMN. The study consists of a double-blinded part A (empasiprubart, IVIg) and an open-label part B (empasiprubart). The maximum study duration for participants is up to 49 months.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the local legal age of consent for clinical studies
* Has a confirmed diagnosis of definite or probable MMN at screening according to the EFNS/PNS 2010 guidelines
* Has responded to IVIg in the past 5 years.
* Is receiving IVIg at a treatment interval of once every 2, 3, 4, or 5 weeks, and a dose of 0.4 to 2.0 g/kg body weight per cycle
* Is receiving a maintenance regimen (no change in frequency, and no change in dose >10%) of IVIg for at least 8 weeks before screening (or at least 10 weeks for participants receiving IVIg once every 5 weeks)
* Minimum converted weekly IVIg dose of ≥0.125 g/kg
* Has documented immunization against encapsulated bacterial pathogens (N meningitidis and S pneumoniae) within 5 years of screening or is willing to receive immunization at least 14 days before first study drug administration

Exclusion Criteria:

* Besides the indication under study, known autoimmune disease (eg, SLE) or any other medical condition that would confound the study results or put the participant at undue risk
* Clinical signs or symptoms suggestive of neuropathies other than MMN, such as motor neuron disease (eg, bulbar signs, brisk reflexes) or other inflammatory neuropathies (eg, sensory neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in grip strength (3-day moving average) in the most affected hand at week 24 | Up to 24 weeks

SECONDARY OUTCOMES:
Change from baseline in MMN-RODS centile score at week 24 | Up to 24 weeks
  The 25-Item Rasch-Built Overall Disability Scale for MMN (MMN-RODS) is a questionnaire about the relationship between daily activities and the participants' health
Change from baseline in mMRC-14 sum score | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
  The modified Medical Research Council (mMRC)-14 is a questionnaire where each muscle group is scored from 0 (paralysis) to 5 (normal strength). A higher value indicates better muscle strength. The total score is based on the sum of both the left and right side of the body.
PGI-C actual value | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
  The Patient Global Impression of Change (PGI-C) is a 7-point scale depicting a participant's rating of overall improvement. The lower the score, the better the improvement.
Change from baseline in CAP-PRI total score | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
  The Chronic Acquired Polyneuropathy Patient-Reported Index (CAP-PRI) includes the assessment of 15 items. Items will be scored 0 (not at all), 1 (a little bit), or 2 (a lot), yielding a total score that ranges from 0 to 30.
Percentage change from baseline in time to complete the 9-HPT with the dominant hand | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
  The 9-Hole Peg Test (9-HPT) is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and nondominant hands will be tested twice (2 consecutive trials of the dominant hand, followed immediately by 2 consecutive trials of the nondominant hand).
Incidence of AEs, AESIs and SAEs | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Serum concentrations over time of empasiprubart | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Percent changes from baseline in free C2 and total C2 over time | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Incidence of anti-drug antibodies (ADA) against empasiprubart in serum | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Incidence of NAb against empasiprubart in serum | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Change from baseline in grip strength (3-day moving average) of the least affected hand over time | Up to 24 weeks
AUC of change from baseline in grip strength (3-day moving average) for the most and least affected hands | Up to 24 weeks
Percentage change from baseline in time to complete the 9-HPT with the nondominant hand over time | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
  The 9-Hole Peg Test (9-HPT) is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and nondominant hands will be tested twice (2 consecutive trials of the dominant hand, followed immediately by 2 consecutive trials of the nondominant hand).
Change from baseline in sum scores for mMRC-10 and mMRC-14 restricted to the 2 most affected muscle groups over time | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
  The modified Medical Research Council (mMRC) is a questionnaire where each muscle group is scored from 0 (paralysis) to 5 (normal strength). A higher value indicates better muscle strength. The total score is based on the sum of both the left and right side of the body.
Proportion of participants and shift from baseline over time by level of severity on PGI-S | Up to 24 weeks
  Patient Global Impression of Severity (PGIS) is a 7-point scale depicting a participant's rating of overall illness severity. Higher scores mean a higher severity.
Change from baseline in Rasch-Transformed Fatigue Severity Scale (RT-FSS) score over time | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Change from baseline in physical component and mental component scores of 12-Item Short Form Survey (SF-12) over time | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Proportion of participants and shift from baseline by each dimension of the EQ-5D-5L scale | Up to 24 weeks (Part A), Up to 120 weeks (Part B)
Changes from baseline in MMN-RODS centile score | Up to 120 weeks (part B)
  The 25-Item Rasch-Built Overall Disability Scale for MMN (MMN-RODS) is a questionnaire about the relationship between daily activities and the participants' health
Changes from baseline in grip strength (3-day moving average; both hands) | Up to 120 weeks (part B)
Actual values of PGI-S over time | Up to 120 weeks (part B)
  Patient Global Impression of Severity (PGIS) is a 7-point scale depicting a participant's rating of overall illness severity. Higher scores mean a higher severity.

CONTACTS AND LOCATIONS:
Locations (102):
- United States (24):
  - HonorHealth Neurology - Bob Bove Neuroscience Institute - Neurology, Scottsdale, Arizona
  - The Neurology Group, Pomona, California
  - Samir Macwan, M.D., Inc., Rancho Mirage, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado - Anschutz Cancer Pavilion (Neuro Onc Clinic), Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - EZR Research LLC, Boca Raton, Florida
  - Healthcare Innovations Institute, LLC, Coral Springs, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Fairway, Kansas
  - Perelman Center for Advanced Medicine, Columbia, Maryland
  - UC Irvine - MDA ALS and Neuromuscular Center, Columbia, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Dent Neurologic Institute Amherst, Amherst, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Morrisville, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - National Neuromuscular Research Institute, Austin, Texas
  - NeuroCarePlus, Houston, Texas
- Australia (4):
  - Royal Melbourne Hospital, Parkville
  - Gold Coast University Hospital, Southport
  - Brain and Mind Center, Sydney
  - Princess Alexandra Hospital, Woolloongabba
- Universitätsklinikum AKH Wien, Vienna, Austria
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Hôpital de la Citadelle, Liège
- Brazil (2):
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto
  - PSEG Centro de Pesquisa Clínica, São Paulo
- Canada (2):
  - Neuro-Outaouais Clinic, Gatineau
  - London Health Sciences Centre, London
- Huashan Hospital Fudan University, Shanghai, China
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet-Inge Lehmanns Vej 8, Copenhagen
- France (10):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU de Brest - Hôpital La Cavale Blanche, Brest
  - Hospices Civils de Lyon - Hôpital Pierre Wertheimer, Bron
  - AP-HP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Roger Salengro, Lille
  - CHU Limoges - Dupuytren 1, Limoges
  - AP-HM- Hôpital de La Timone, Marseille
  - CHU de Nice-Hôpital Pasteur, Nice
  - AP-HP - Hôpital de la Pitié Salpétrière, Paris
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
- Germany (6):
  - Universitätsklinikum Essen, Essen
  - Universität Georg August, Göttingen
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Universitätsklinikum Münster, Münster
  - Alexianer - MVZ St. Josefs-Krankenhaus Potsdam GmbH, Potsdam
  - Universitätsklinikum Würzburg, Würzburg
- Greece (2):
  - University General Hospital ''ATTIKON'' - General Hospital of West Attica H AGIA VARVARA, Chaïdári
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
- Italy (8):
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Fondazione Serena Onlus - Centro Clinico NeMO Brescia, Gussago
  - Az. Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Milan
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Japan (6):
  - Juntendo University Hospital, Bunkyō City
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Chiba University Hospital, Chūōku
  - National Center of Neurology and Psychiatry, Kodaira
  - Nagoya University Hospital, Nagoya
  - Yamaguchi University Hospital, Ube
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania
- Amsterdam UMC, Amsterdam, Netherlands
- Oslo Universitetssykehus HF, Ullevål, Oslo, Norway
- Poland (5):
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Neurologia Slaska, Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Galen Clinic -- Lublin, Lublin
  - UCK WUM, Centralny Szpital Kliniczny, Warsaw
- ULS de Santo António, EPE - Hospital de Santo António, Porto, Portugal
- University Clinical Center of Serbia, Belgrade, Serbia
- Slovakia (2):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Univerzitna nemocnica MARTIN, Martin
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (9):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Basurto, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Universitario de Donostia, San Sebastián
- Inselspital - Universitätsspital Bern, Bern, Switzerland
- United Kingdom (4):
  - Queen Elizabeth University Hospital, Glasgow
  - John Radcliffe Hospital, Oxford
  - Salford Royal Hospital, Salford
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No